CLINICAL TRIAL: NCT00465088
Title: SUPREME: A 12-Week, Open-Label, Multicenter Study to Compare the Lipid Effects of Niacin ER and Simvastatin (NS) to Atorvastatin in Subjects With Hyperlipidemia or Mixed Dyslipidemia
Brief Title: An Open-Label Study to Compare the Lipid Effects of Niacin ER and Simvastatin (NS) to Atorvastatin in Subjects With Hyperlipidemia or Mixed Dyslipidemia (SUPREME)
Acronym: SUPREME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Scott Krause, AD Clinical Research, Abbott
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 019-05-06-CR; M10-013
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Results first posted 2009-05-13 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Hyperlipidemia; Mixed Dyslipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Simcor; Atorvastatin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Niacin ER/Simvastatin Tablets
- 2 (Experimental)
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: Niacin ER/Simvastatin Tablets — Up to 2000 mg/40 mg at bedtime
  Other Names: ABT-919/483; Niacin ER/Simvastatin; Simcor
  Arms: 1
Drug: atorvastatin — 40 mg at bedtime
  Arms: 2

SUMMARY:
To demonstrate that niacin ER and simvastatin (NS) tablets, when compared to atorvastatin (Lipitor®; Pfizer, Inc.), has superior high-density lipoprotein cholesterol (HDL-C) elevating effects at Week 12 in subjects with type II hyperlipidemia or mixed dyslipidemia who are currently off lipid-modifying therapy. This was a prospective, randomized, open-label, blinded endpoint (PROBE) study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following laboratory criteria:

  * HDL-C <40 mg/dL for men and <50 mg/dL for women.
  * LDL-C ≥130 mg/dL but <250 mg/dL.
  * TG <350 mg/dL.
  * Creatine phosphokinase (CPK) < 3 x upper limit of normal (ULN).
  * Alanine aminotransferase (ALT); serum glutamic pyruvic transaminase [SGPT] and aspartate aminotransferase (AST); serum glutamic oxaloacetic transaminase [SGOT] < 1.3 x ULN.
* Subjects must also be reasonably compliant with the Therapeutic Lifestyle Changes (TLC) diet during the 4 to 5 week Screening Period prior to randomization (and be willing to comply for the duration of the study).

Exclusion Criteria:

* Subjects who have a history of any important medical conditions or abnormalities (as specified in the protocol) that would preclude study inclusion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Thakkar, MD, Study Director — Abbott
Locations (46):
- United States (46):
  - Anaheim, California
  - Huntington Park, California
  - Long Beach, California
  - Sacramento, California
  - Walnut Creek, California
  - Brooksville, Florida
  - Daytona Beach, Florida
  - Gainesville, Florida
  - Largo, Florida
  - Merritt Island, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Calhoun, Georgia
  - Decatur, Georgia
  - Dunwoody, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Arkansas City, Kansas
  - Newton, Kansas
  - Shawnee Mission, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Auburn, Maine
  - Baltimore, Maryland
  - Missoula, Montana
  - Charlotte, North Carolina
  - High Point, North Carolina
  - Canfield, Ohio
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Protland, Oregon
  - Chicora, Pennsylvania
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Austin, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Magna, Utah
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Gig Harbor, Washington
  - Menomonee Falls, Wisconsin
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 199 subjects randomized, 6 did not receive study drug: 2 withdrew consent, 1 had a protocol violation, and 3 had randomization errors. 193 subjects were treated.
Groups:
- Niacin Extended-release Plus Simvastatin: Up to 2000 mg of niacin extended-release plus 40 mg simvastatin once daily at bedtime
- Atorvastatin: 40 mg atorvastatin once daily at bedtime
Period: Overall Study
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Started | 114 (For both arms, started means treated.) | 79
Completed | 82 | 70
Not Completed | 32 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin | Total
Number analyzed (Participants) | 114 | 79 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 73 | 166
  >=65 years | 21 | 6 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 55.1 (12.06) | 51.5 (11.12) | 53.6 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 38 | 109
  Male | 43 | 41 | 84
Region of Enrollment [Number; unit: participants]
  United States | 114 | 79 | 193

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 12
Description: (Week 12 HDL-C minus baseline HDL-C) x 100/baseline HDL-C
Time Frame: From baseline to Week 12
Population: All treated subjects whose Week 12 value was obtained within the Week 12 visit window
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 82 | 70
percent change | 30.1 [25.6 to 34.6] | 9.4 [4.3 to 14.4]
Statistical Analysis 1: Comparison: Niacin Extended-release Plus Simvastatin vs Atorvastatin; An n = 81 for niacin extended-release with simvastatin and n = 54 for atorvastatin would provide > 99% power to detect a 13% increase in HDL-C with niacin extended-release with simvastatin relative to atorvastatin, assuming an SD of 16%; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — alpha = 0.05

2. Secondary Outcome: Percent Change in HDL-C From Baseline to Week 8
Description: (Week 8 HDL-C minus baseline HDL-C) x 100/baseline HDL-C
Time Frame: From baseline to Week 8
Population: All treated subjects whose Week 8 value was obtained within the Week 8 visit window
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 85 | 72
percent change | 26.7 [23.1 to 30.2] | 1.4 [-2.7 to 5.4]

3. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Week 8
Description: (Week 8 non-HDL-C minus baseline non-HDL-C) x 100/baseline non-HDL-C
Time Frame: From baseline to Week 8
Population: All treated subjects whose Week 8 value was obtained within the Week 8 visit window
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 85 | 70
percent change | -45.0 [-48.9 to -41.0] | -44.3 [-48.8 to -39.8]

4. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Week 12
Description: (Week 12 non-HDL-C minus baseline non-HDL-C) x 100/baseline non-HDL-C
Time Frame: From baseline to Week 12
Population: All treated subjects whose Week 12 value was obtained within the Week 12 visit window
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 82 | 70
percent change | -43.4 [-47.7 to -39.0] | -43.3 [-48.2 to -38.5]

5. Secondary Outcome: Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 12
Description: (Week 12 LDL-C minus baseline LDL-C) x 100/baseline LDL-C
Time Frame: From baseline to Week 12
Population: All treated subjects whose Week 12 value was obtained within the Week 12 visit window (between 70 days after first dose and not more than 3 days after last dose)
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 82 | 70
percent change | -43.8 [-48.3 to -39.2] | -46.0 [-51.0 to -40.9]

6. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 12
Description: (Week 12 triglycerides minus baseline triglycerides) x 100/baseline triglycerides
Time Frame: From baseline to Week 12
Population: All treated subjects whose Week 12 value was obtained within the Week 12 visit window
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 82 | 70
percent change | -44.0 [-62.8 to -20.9] | -37.0 [-47.8 to -18.8]

7. Secondary Outcome: Percent Change in LDL-C:HDL-C Ratio
Description: (Week 12 LDL-C:HDL-C ratio minus baseline LDL-C:HDL-C ratio) x 100/baseline LDL-C:HDL-C ratio
Time Frame: From baseline to Week 12
Population: All treated subjects whose Week 12 values were obtained within the Week 12 visit window
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 82 | 70
percent change | -54.5 [-59.1 to -49.8] | -50.5 [-55.7 to -45.3]

8. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Week 12
Description: (Week 12 total cholesterol minus baseline total cholesterol) x 100/baseline total cholesterol
Time Frame: From baseline to Week 12
Population: All treated subjects whose Week 12 value was obtained within the Week 12 visit window
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 82 | 70
percent change | -31.3 [-34.8 to -27.7] | -35.1 [-39.1 to -31.1]

9. Secondary Outcome: Percent Change in Total Cholesterol:HDL-C Ratio
Description: (Week 12 total cholesterol:HDL-C ratio minus baseline total cholesterol:HDL-C ratio) x 100/baseline total cholesterol:HDL-C ratio
Time Frame: From baseline to Week 12
Population: All treated subjects whose Week 12 values were obtained within the Week 12 visit window
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 82 | 70
percent change | -45.2 [-49.0 to -41.3] | -40.3 [-44.7 to -36.0]

10. Secondary Outcome: Percent Change in Lipoprotein A From Baseline to Week 12
Description: (Week 12 lipoprotein A minus baseline lipoprotein A) x 100/baseline lipoprotein A
Time Frame: From baseline to Week 12
Population: All treated subjects whose Week 12 value was obtained within the Week 12 visit window
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 82 | 70
percent change | -15.8 [-36.8 to 8.8] | 16.0 [-7.1 to 30.8]

11. Secondary Outcome: Percentage of Subjects Meeting With HDL-C >/= 40 mg/dL at Week 12
Time Frame: 12 weeks
Population: All treated subjects not meeting National Cholesterol Education Program Adult Treatment Panel (NCEP ATP) III goals at baseline with both a baseline and at least 1 postbaseline HDL-C value
Measure: Number; unit: Percentage of subjects
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 45 | 47
Percentage of subjects | 78 | 28

12. Secondary Outcome: Percentage of Subjects Meeting National Cholesterol Education Program Adult Treatment Panel (NCEP ATP) III Goal for LDL-C at Week 12
Description: For high-risk patients (coronary heart disease or equivalent), LDL-C < 100 mg/dL and non-HDL-C < 130 mg/dL; for moderate risk patients (having 2 risk factors), LDL-C < 130 mg/dL and non-HDL-C < 160 mg/dL; for low-risk patients (having 0 or 1 risk factor): LDL-C < 160 mg/dL and non-HDL-C < 190 mg/dL.
Time Frame: 12 weeks
Population: All treated subjects not meeting NCEP ATP III goals at baseline with both a baseline and at least 1 postbaseline LDL-C value
Measure: Number; unit: Percentage of subjects
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 67 | 58
Percentage of subjects | 78 | 84

13. Secondary Outcome: Percentage of Subjects With Triglycerides < 150 mg/dL at Week 12
Time Frame: 12 weeks
Population: All treated subjects not meeting NCEP ATP III goals at baseline with both a baseline and at least 1 postbaseline triglyceride value
Measure: Number; unit: Percentage of subjects
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 52 | 44
Percentage of subjects | 79 | 70

14. Secondary Outcome: Percentage of Subjects With HDL-C >/= 40 mg/dL, LDL-C Meeting NCEP ATP III Goal, and Triglycerides < 150 mg/dL at Week 12
Description: NCEP ATP III goals for LDL-C are as follows: For high-risk patients, LDL-C < 100 mg/dL; for moderate risk patients, LDL-C < 130 mg/dL; for low-risk patients: LDL-C < 160 mg/dL. High-risk means coronary heart disease or risk equivalents; moderate risk means having at least 2 risk factors; low-risk means having no or 1 risk factor.
Time Frame: 12 weeks
Population: All treated subjects not meeting NCEP ATP III goals at baseline with both a baseline and at least 1 postbaseline value for all 3 lipid parameters
Measure: Number; unit: Percentage of subjects
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Number analyzed (Participants) | 79 | 65
Percentage of subjects | 65 | 34

ADVERSE EVENTS:
Arm/Group | Niacin Extended-release Plus Simvastatin | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 2 | 1
Other Adverse Events (participants affected / at risk) | 89 | 27
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Niacin Extended-release Plus Simvastatin | Atorvastatin
Coronary artery disease (Cardiac disorders) | 1/114 | 0/79
Chest pain (General disorders) | 1/114 | 1/79
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Niacin Extended-release Plus Simvastatin | Atorvastatin
Abdominal distension (Gastrointestinal disorders) | 0/114 | 2/79
Constipation (Gastrointestinal disorders) | 5/114 | 0/79
Diarrhea (Gastrointestinal disorders) | 9/114 | 2/79
Nausea (Gastrointestinal disorders) | 9/114 | 0/79
Vomiting (Gastrointestinal disorders) | 11/114 | 0/79
Edema peripheral (General disorders) | 0/114 | 2/79
Nasopharyngitis (Infections and infestations) | 2/114 | 2/79
Tooth infection (Infections and infestations) | 3/114 | 0/79
Joint sprain (Injury, poisoning and procedural complications) | 0/114 | 2/79
Blood creatinine phosphokinase increased (Investigations) | 0/114 | 2/79
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/114 | 2/79
Arthritis (Musculoskeletal and connective tissue disorders) | 0/114 | 2/79
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0/114 | 2/79
Myalgia (Musculoskeletal and connective tissue disorders) | 4/114 | 4/79
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3/114 | 1/79
Dizziness (Musculoskeletal and connective tissue disorders) | 3/114 | 2/79
Headache (Nervous system disorders) | 9/114 | 2/79
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/114 | 2/79
Pruritus (Skin and subcutaneous tissue disorders) | 7/114 | 0/79
Flushing (Vascular disorders) | 77/114 | 8/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to release; Sponsor shall receive up to 180 days for review. Differences shall be resolved in good faith through appropriate scientific debate.